CLINICAL TRIAL: NCT03793933
Title: Performance of the American College of Surgeons Surgical Risk Calculator in Patients Undergoing Hepatectomy for Liver Tumors
Brief Title: ACS-NSQIP Calculator for Liver Surgery
Status: Completed | Type: Observational
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Matteo Donadon, Assistant Professor of Surgery, Humanitas Clinical and Research Center
Other Study IDs: ACS-NSQIP
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Liver Surgery; Hepatectomy; Outcome After Hepatectomy
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Liver resection — Surgery for the liver
  Other Names: Hepatectomy

SUMMARY:
The American College of Surgeons National Surgical Quality Improvement Program's (ACS-NSQIP) calculator has been endorsed by the surgeons' community to counsel patients and relatives regarding estimated postoperative complications. However, it does not include organ-specific risks. The aim of this study was to assess the ACS-NSQIP calculator's ability to predict complications, mortality and length of stay (LOS) in patients undergoing hepatectomy for liver tumors

DETAILED DESCRIPTION:
This is an observational retrospective study conducted in a tertiary-referral university hospital. An established classification of complications, including post-hepatectomy insufficiency and bile leak, was adopted. The endpoint was the rate of complications, mortality and LOS as expected by the ACS-NSQIP calculator and as observed within 90-day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who underwent surgery for a liver tumor at our Institution between the defined period of time

Exclusion Criteria:

* Any patient with missing data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study examined a cohort of consecutive patients that underwent hepatectomy at our institution between November 2015 and July 2018.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
ACS-NSQIP calculator's ability | From the date of surgery up to three months from the date of surgery
  The primary study endpoint was to assess the ACS-NSQIP calculator's ability to predict complications, mortality and length of stay in patients undergoing hepatectomy for liver tumors

IPD SHARING:
Plan to Share IPD: No